CLINICAL TRIAL: NCT05164835
Title: Study of Drug Acceptance and Its Persistence Over Time in Patients Receiving a Haematopoietic Stem Cell Allograft: a Pilot Study at the University Hospital of Limoges
Brief Title: Study of Drug Acceptance and Its Persistence Over Time in Patients Receiving a Haematopoietic Stem Cell Allograft
Acronym: AdHemLim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 87RI21_0032 (AdHemLim)
Record Dates: First submitted 2021-10-31; First posted 2021-12-21 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-01

CONDITIONS: Allograft
Keywords: allograft; drug; acceptance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: pharmaceutical follow-up

INTERVENTIONS:
Other: pharmaceutical follow-up — Pharmaceutical follow-up over 1 year and pharmaceutical interviews during the various medical consultation appointments.
  In addition to the usual care:
  * Delivery of questionnaire at the time defined in the protocol. The questionnaires will be given during the waiting time of the patients at the University Hospital of Limoges.
  * Extension of the duration of the usual interview by 10 minutes in order to collect the desired information.

SUMMARY:
Allograft patients have a complex care pathway and are left with a large number of prescribed medications.

They have to deal with changes linked to the transplant (change in taste, fatigue, regular monitoring, risk of GVH (graft versus host) complications, infectious risks, change in eating habits, etc.), and a large number of associated drugs (immunosuppressants, anti-infectious prophylaxis and supplements (folic acid, magnesium, bile salts, etc.), which are added to any pre-existing chronic pathologies.

Therapeutic adherence of these patients is a real challenge. Indeed, the success of the transplant and the complications that may arise (graft rejection, GVH, infections, death, hospitalisation, etc.) are closely linked to good or poor therapeutic adherence. Moreover, the majority of these patients are young and are not used to taking many treatments, which will change after the transplant.

Adherence to treatment consists of three phases:

* Acceptance of the disease and the benefits of treatment,
* Compliance: following the instructions of the prescription (dosage and schedule),
* Persistence: consistency of compliance over time.

Support from the care team throughout the management of these patients is necessary for good therapeutic adherence in order to prevent and act early on the difficulties encountered (appearance of side effects linked to the treatments, large number of tablets per day, duration of treatment (1 to 2 years), risk of GVH, significant asthenia and difficulty in concentrating, etc.)

We have a large amount of data on therapeutic adherence and potential non-adherence factors in patients with chronic diseases (diabetes, asthma, cancer, etc.) or in solid organ transplant patients.

On the other hand, there is little data on allograft patients. Most often, a parallel is made between the data present in kidney transplant patients and allograft patients. However, it is necessary to study more specifically the therapeutic adherence in this population.

A recent multicentre cross-sectional study in France on adherence in allograft patients showed that 80% of adult and paediatric patients were not adherent.

ELIGIBILITY:
Inclusion Criteria:

* allograft patients followed by the Limoges University Hospital

Exclusion Criteria:

* patient hospitalised at the Limoges University Hospital for a reason other than allograft
* refusal of the patient to participate in this research
* patient unable to understand the treatment
* pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Medication adherence level | month 12
  Patient's level of medication adherence will be assessed by the 8-item Morisky test (score 0 to 13 : a score greater than or equal to 11 show good adherence)
Factors associated with a change | month 12
  Semi-structured interview conducted at M+12 post-transplant.

SECONDARY OUTCOMES:
Medication adherence level | day 15
  Patient's level of medication adherence will be assessed by the 8-item Morisky test (score 0 to 13 : a score greater than or equal to 11 show good adherence)
Factors associated with a change | day 15
  Semi-structured interview conducted at D+15 after discharge from hospital.
Medication adherence level | month 3
  Patient's level of medication adherence will be assessed by the 8-item Morisky test (score 0 to 13 : a score greater than or equal to 11 show good adherence)
Factors associated with a change | month 3
  Semi-structured interview conducted at M+3 post-transplant.
Medication adherence level | month 6
  Patient's level of medication adherence will be assessed by the 8-item Morisky test (score 0 to 13 : a score greater than or equal to 11 show good adherence)
Factors associated with a change | month 6
  Semi-structured interview conducted at M+6 post-transplant.
Medication adherence level | month 9
  Patient's level of medication adherence will be assessed by the 8-item Morisky test (score 0 to 13 : a score greater than or equal to 11 show good adherence)
Factors associated with a change | month 9
  Semi-structured interview conducted at M+9 post-transplant.
Patient's representations of their medication after transplantation | day 15
  Use of the "belief about medicines" questionnaire : 18 items. Each item is rated from 0 to 5 (0 = strongly disagree, 5 = strongly agree)
Patient's representations of their medication after transplantation | day 15
  semi-directive interview approach using specific items
Patient's representations of their medication after transplantation | month 6
  Use of the "belief about medicines" questionnaire : 18 items. Each item is rated from 0 to 5 (0 = strongly disagree, 5 = strongly agree)
Patient's representations of their medication after transplantation | month 6
  semi-directive interview approach using specific items
Patient's representations of their medication after transplantation | month 12
  Use of the "belief about medicines" questionnaire : 18 items. Each item is rated from 0 to 5 (0 = strongly disagree, 5 = strongly agree)
Patient's representations of their medication after transplantation | month 12
  semi-directive interview approach using specific items
Representation of the information given on transplant drugs according to the health professionals accompanying the transplant patient | day 0
  ad hoc closed-ended questionnaire conducted prior to transplantation
Representation of the information given on transplant drugs according to the health professionals accompanying the transplant patient | month 3
  ad hoc closed-ended questionnaire
Representation of the information given on transplant drugs according to the health professionals accompanying the transplant patient | month 6
  ad hoc closed-ended questionnaire
Representation of the information given on transplant drugs according to the health professionals accompanying the transplant patient | month 12
  ad hoc closed-ended questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No